CLINICAL TRIAL: NCT05533151
Title: The Influence of Telerehabilitation Focused on Respiratory Muscle Training on the Functional Status of Patients With the Respiratory System Diseases
Brief Title: The Influence of Telerehabilitation Focused on Respiratory Muscle Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Zdenek Svoboda, Assoc. Prof. Zdenek Svoboda, Ph.D., Palacky University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSGC-2021-0156
Record Dates: First submitted 2022-07-25; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Telerehabilitation
Keywords: Respiratory muscle training; Pulmonary rehabilitation; Telerehabilitation; Respiratory system disease; Physical activity; Functional status; Exercise tolerance; Spirometry
MeSH Terms: conditions — Respiratory Tract Diseases; Motor Activity | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: All study participants will be divided into 3 groups according to their lung disease. Each group should contain 20 patients, who will be randomly split into an intervention and a control group of 10 patients each.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bronchial asthma (Experimental): This group envolves parients suffering from bronchial asthma.
  Interventions: Device: Respiratory muscle training
- Interstitial lung diseases (Experimental): This group envolves parients suffering from interstitial lung disease.
  Interventions: Device: Respiratory muscle training
- Lung transplantation (Experimental): This group envolves parients after lung transplantation done for a pulmonary disease.
  Interventions: Device: Respiratory muscle training

INTERVENTIONS:
Device: Respiratory muscle training — All patients will be initially educated by a physiotherapist and instructed to independently perform the home exercise program including respiratory muscle training. The training will be performed using the Airofit PRO device. This breathing training on a suitable resistance will be performed twice a day for 6 weeks. The intervention will be conducted under a researcher's supervision via smartphone App.

SUMMARY:
Pulmonary rehabilitation, which includes respiratory muscle training, is effective in improving the functional status of patients with various types of the respiratory system diseases, including bronchial asthma, interstitial lung diseases or lung transplant patients.

However, availability of pulmonary rehabilitation is limited in the Czech Republic. Nowadays even more due to the Covid-19 pandemic. A suitable instrument of increasing its accessibility is telerehabilitation using modern technologies. The main goal of this project is to evaluate the patients' functional status after completing a standardized cycle of pulmonary rehabilitation focused on respiratory muscle training conducted as telerehabilitation sessions and compare the effect of this intervention with a different group of patients who will undergo an education session led by a trained physiotherapist followed by self-directed exercise according to an exercise brochure.

DETAILED DESCRIPTION:
The study will include patients with the following respiratory system diseases: bronchial asthma, interstitial lung diseases (sarcoidosis, pulmonary fibrosis, etc.) and patients after lung transplantation enrolled in outpatient care by the attending physician.

All these patients must meet inclusion criteria, such as: stable disease status, no exacerbation within last 2 months. Patients with comorbidities (rheumatological, neurological, psychiatric, etc.) preventing them from being enrolled in a pulmonary rehabilitation program will be excluded from the study. All study participants will be divided into 3 groups according to their lung disease. Each group should contain 20 patients, who will be randomly split into an intervention and a control group of 10 patients each. The course of lung disease, its symptoms, medication, and the patient's functional status will be determined in detail. The following parameters will be objectively evaluated: lung function and respiratory muscle strength, exercise tolerance, chest expansion, dyspnoea, fatigue, anxiety and depression, quality of life in relation to lung disease and physical activity. The patients will be examined using spirometry, Modified Medical Research Council Dyspnea Scale, the Multidimensional Assessment of Fatigue Scale, self-report Beck Depression Inventory-II scale for adults and St. George's Respiratory Questionnaire examining the quality of life in relation to lung disease. Exercise tolerance testing will be performed through a 1-minute Sit-to-stand test. The level of physical activity will be examined using Axivity AX3 accelerometers, which the patient will wear for 7 days after the initial assessment, which will take place in one day. There will always be a long enough rest between examinations, so that fatigue cannot affect the course of the measurement. All assessments are non-invasive, and all the mentioned test methods are standardized and commonly used in patients with diseases of the respiratory system according to the recommendations of the Czech Pneumological and Phthisiological Society and the European Respiratory Society. All patients will be initially educated by a physiotherapist and instructed to independently perform the home exercise program including respiratory muscle training. This program will also include breathing exercises to correct the breathing pattern, exercises to strengthen the upper and lower limbs muscles, balance exercises and recommendations for endurance training. Respiratory muscle training will be performed using the Airofit PRO device. This breathing device can be set to a suitable resistance for both inhale and exhale to increase the strength of the inspiratory and expiratory muscles. Airofit PRO device can also be connected to an application in a smartphone, which records the ongoing results of the training as well as the frequency of the device use. This is a great starting point for its implementation within a telerehabilitation program, as well as for its self-directed use. The intervention group will perform the home exercise program independently with the use of an exercise brochure and at the same time with the support of telerehabilitation lessons with a physiotherapist twice a week via Zoom meeting. The control group will continue in a separate program according to the exercise brochure. To ensure a correct exercise performance all exercises in the exercise brochure will be individually practiced by a trained physiotherapist with each patient from both groups during the initial assessment. The assessment day will be divided into two parts:

1. all assessments in the morning; 2. exercise brochure introduction in the afternoon to avoid fatigue of patients. The final assessment will take place 6 weeks after the initial one. It will be exactly the same as the first one.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bronchial asthma
* diagnosis of interstitial lung disease
* post-lung-transplantation statust
* stable disease status
* no exacerbation within last 2 months.

Exclusion Criteria:

* serious comorbidities (rheumatological, neurological, psychiatric, etc.)
* other respiratory lung disease than the specified ones
* contraindication for respiratory muscle training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | 6 weeks
  Respiratory muscle strength (MIP = maximum inspiratory pressure, MEP = maximum expiratory pressure, P0.1 = airway occlusion pressure [kPa], TTmus = tension time index). Evaluation of the difference between respiraory muscle strength training with (intervention) and without (control) telerehabilitation support.
The adherence to respiratory muscle training | 6 weeks
  The frequency (number) of the smartphone App use is the main determinant for the adherence evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Raisova, Assoc.Prof., Study Director — Palacký University, Olomouc
Locations (1):
- Faculty of Physical Culture, Palacky University Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No